CLINICAL TRIAL: NCT04252677
Title: Health Literacy as a Vehicle to Reduce Obesogenic Behaviors Among Adolescents: A Pilot Intervention
Brief Title: Health Literacy and Obesogenic Behaviors
Acronym: HL-Squared
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City University of New York, School of Public Health (Other)
Responsible Party: Principal Investigator, Sasha Fleary, Associate Professor, City University of New York, School of Public Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HLSQUARED01
Record Dates: First submitted 2020-01-16; First posted 2020-02-05 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Obesity, Adolescent; Health Behavior; Health Knowledge, Attitudes, Practice; Diet, Healthy; Exercise; Health Literacy
Keywords: health literacy; obesity; diet; physical activity; information-motivation-behavioral skills model; adolescent
MeSH Terms: conditions — Pediatric Obesity; Health Behavior; Behavior; Motor Activity; Obesity | interventions — Health Literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaping and Obesity Prevention Only (Active Comparator): Obesity prevention and vaping
  1. Vaping:
     * Factual information about vaping devices and vaping
     * Beliefs and attitudes about nicotine products
     * Refusing and avoiding vaping
     * Recognizing addiction and getting help
  2. Health information:
     • Factual information about healthy eating and activity (PA)
  3. Motivation:
     * Personal: Create positive attitudes toward engagement in healthy eating and PA
     * Social: Enlisting social support to increase healthy eating and PA
     * Social: Identification of community resources that promote and support healthy eating and PA
  4. Behavioral Skills
     * Tips for engaging in prevention behaviors and avoiding risk behaviors in the context of existing barriers
     * Skills for social situations around behaviors
     * Skills for making behavior part of routine
     * Build autonomy, self-efficacy and model good health decision-making for health behaviors
  Interventions: Behavioral: Obesity Prevention
- Health Literacy and Obesity Prevention (Experimental): Obesity prevention and health literacy (HL).
  1. Health Literacy
     * Functional HL: skills for reading/understanding nutrition labels and medication instructions.
     * Interactive HL: verbal skills for interacting with others on health issues.
     * Critical HL: connections between advocacy and health
     * Media HL: skills for accessing and identifying reliable source of media.
  2. Health information:
     • Factual information about healthy eating and activity (PA)
  3. Motivation:
     * Create positive attitudes toward engagement in healthy eating and PA
     * Enlisting social support to increase healthy eating and PA
     * Identification of community resources that promote and support healthy eating and PA
  4. Behavioral Skills
     * Tips for engaging in prevention behaviors and avoiding risk behaviors
     * Skills for social situations around behaviors
     * Skills for making behavior part of routine
     * Build autonomy, self-efficacy and good health decision-making for health behaviors
  Interventions: Behavioral: Obesity Prevention; Behavioral: Health Literacy

INTERVENTIONS:
Behavioral: Obesity Prevention — This intervention includes content specific to obesity behaviors-related health information, motivation, and behavioral skills.
Behavioral: Health Literacy — This intervention includes content specific to improving health literacy.
  Arms: Health Literacy and Obesity Prevention

SUMMARY:
The prevalence of adolescent behaviors that can lead to obesity are alarming, and reduced life expectancy is the future of America's youth if behavioral changes are not implemented to improve health and reduce the obesity burden. Researchers have argued that health literacy is a precursor to health knowledge and is necessary for translating knowledge about healthy choices into behavior, with low health literacy being associated with reduced preventive health behaviors in adults. Given the lack of health literacy-specific interventions addressing adolescents' obesogenic behaviors, the purpose of this study is to examine the preliminary effectiveness of adding a health literacy module to an obesity prevention intervention that addresses adolescents' obesogenic behaviors.

DETAILED DESCRIPTION:
The rates of pediatric obesity (~19%) and diabetes (0.24%) in the US are alarming and behaviors implicated in obesity and type 2 diabetes are highly prevalent. Approximately 69% and 73% of adolescents consume less than two fruits and vegetables daily respectively, while 53% engage in insufficient physical activity. These behaviors magnify adolescents' immediate and long-term risks for obesity and obesity-related chronic illnesses, as well as complicate the treatment of obesity-related chronic illnesses. Children and adolescents who are obese are four times more likely to be diagnosed with type 2 diabetes than normal weight children, with serious short and long-term consequences impacting quality of life. Reduced life expectancy is the future of America's youth if behavioral changes are not implemented to improve health and reduce the obesity burden. Reversing current national trends in obesity and type 2 diabetes require novel and sustainable prevention strategies to address children and adolescents' obesogenic behaviors.

Adolescence is marked by increased autonomy in decision-making, yet data suggest that adolescents are not equipped with all the skills to make effective health-related behavioral decisions. While health knowledge works in conjunction with motivation and behavioral skills to predict behavior, most existing adolescent interventions target these variables in isolation with modest success. Researchers have argued that health literacy (HL) - the ability to access, understand, and use health information to make informed health decisions - is a precursor to health knowledge and is necessary for translating health knowledge into behavior. Low HL among adults is associated with poor ability to interpret health messages, and results in reduced preventive health behaviors. Further, parent and adolescent HL is negatively related to adolescents' obesity status. Thus, while research on adding HL to existing behavior interventions to improve adolescents' obesity prevention behaviors is lacking, it is expected that the inclusion of HL into existing interventions will increase intervention effectiveness and positive behavior outcomes.

The long-term goal of this line of research is to reduce the incidence of obesity in adolescents and by extension reduce the risk for obesity-related chronic illnesses using interventions that address individual and contextual factors related to long-term health decision-making and behavior change. The goal of the proposed study is to examine the effect of adding a HL component to an obesity prevention intervention that addresses adolescents' obesogenic behavior-related health knowledge, motivation, and behavioral skills. The central hypothesis is adolescents receiving HL training as part of an obesity prevention intervention will have higher rates of prevention behaviors than those in the obesity prevention only condition. Study goals will be achieved through the following specific aims:

Aim 1: Modify successful components of existing obesity prevention interventions into an interactive digital platform with and without HL for acceptability and usability in adolescents.

Approach: Use successful components of existing interventions, our completed preliminary research, and our research teams' expertise to develop an interactive digital intervention including HL, and obesogenic behavior-related health knowledge, motivation, and behavioral skills. Assess and modify the intervention for usability and acceptability among 14-16-year-olds through an iterative process.

Aim 2: Determine if the addition of HL training to an interactive digital obesity prevention intervention will improve adolescents' obesity prevention behaviors over the obesity intervention alone.

Hypothesis: Adolescents in the obesity prevention plus HL intervention will have higher rates of obesity prevention behaviors at posttest and follow-up compared to the obesity prevention only group.

Approach: Conduct a two-arm randomized controlled trial (RCT) intervention (obesity prevention only, obesity prevention/HL) and estimate the intervention's effects on obesogenic behaviors. Adolescents (n = 76; 14-16-year-olds) will be randomly assigned to each condition (38/condition). Conduct pretest, posttest, and 1- and 3-month assessments of HL, obesogenic behaviors, and obesogenic behavior-related motivation, behavioral skills, and knowledge.

Outcomes: Intervention completion will result in effect size estimates of improvements in obesity prevention behaviors, health knowledge, motivation, and behavioral skills for both groups with greater improvements for the HL group at posttest and follow-up. The obesity prevention/HL intervention group will also have higher HL at posttest and follow-up. Retention, recruitment, completion and treatment fidelity rates will be established.

Innovation & Impact: This study incorporates HL, an understudied but potentially critical factor in adolescents' health behaviors. The intervention will be developed and implemented in a digital format which will increase reach and impact. This is the first study examining the effect of including HL in adolescents' obesity prevention interventions. This study sets the groundwork for a full scale, RCT to assess the benefit of HL training added to an obesity prevention intervention to address adolescents' obesogenic behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents 13-16 years old at time of enrollment (may turn age 17 during the study
* Must have parental consent
* All weight classifications

Exclusion Criteria:

* Adolescents younger than 13 years or older than 16 years at time of enrollment
* No parental consent
* Medical conditions preventing engagement in physical activity
* Medical conditions resulting in extremely restricted diets (e.g., ketogenic diet)
* Already participating in an intervention related to healthy eating, physical activity and/or obesity prevention or treatment

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Improvement in participants' healthy eating behaviors as assessed by the Dietary Screener Questionnaire | 5 months
  Recall of healthy eating (e.g., fruits and vegetables, whole grain, fiber, calcium) behaviors
Reductions in participants' unhealthy eating behaviors as assessed by the Dietary Screener Questionnaire | 5 months
  Recall of unhealthy eating (sugary and salty foods, fast foods, sugar-sweetened beverages, saturated fats) behaviors
Improvement in participants' healthy eating behaviors as assessed by the National Youth Physical Activity and Nutrition Study | 5 months
  Recall of healthy eating (e.g., fruits and vegetables, whole grain, fiber, calcium) behaviors
Reductions in participants' unhealthy eating behaviors as assessed by the National Youth Physical Activity and Nutrition Study | 5 months
  Recall of unhealthy eating (sugary and salty foods, fast foods, sugar-sweetened beverages, saturated fats) behaviors
Improvements in participants' physical activity as assessed by the Youth Activity Profile | 5 months
  Recall of moderate and vigorous physical activity behaviors
Improvements in participants' physical activity as assessed by the Godin and Shephard Leisure-Time Physical Activity Questionnaire | 5 months
  Recall of moderate and vigorous physical activity behaviors
Reductions in participants' sedentary activity as assessed by the Youth Activity Profile | 5 months
  Recall of sedentary activity behaviors

SECONDARY OUTCOMES:
Participants' functional health literacy will be assessed using the Newest Vital Signs | 5 months
  Objective measure of reading and numeracy skills for health
Participants' interactive and critical health literacy will be assessed using the Assesments of Adolescent Health Literacy Scales | 5 months
  Objective measure of social skills and critical thinking for health
Participants' media health literacy will be measured using the Adolescent Media Health Literacy Scale and eHeals | 5 months
  Measures of media literacy for health
Participants' physical activity knowledge will be assessed using the knowledge and understanding subscale of the Canadian Assessment of Physical Literacy | 5 months
  Measures awareness of fitness terminology, physical and sedentary activity recommendations, and use of safety equipment during physical activity
Participants' nutrition knowledge will be assessed using a modified General Nutrition Knowledge Questionnaire for Adults | 5 months
  Measures knowledge of dietary recommendations, sources of nutrients, choosing everyday foods and diet-disease relationships
Participants' personal motivation will be assessed using the Regulation of Eating Behaviors Scale | 5 months
  Assesses autonomous motivation, controlled motivation, and amotivation for diet and physical activity
Participants' social motivation for diet will be assessed using the decisional balance, family influences, and peer influences subscales of the Psychosocial Constructs for Adolescent Fruit and Vegetables and Dietary Fat Intake Questionnaire | 5 months
  Social motivation will be assessed using the decisional balance, family influences, and peer influences subscales
Participants' social motivation for physical activity will be assessed using the decisional balance, family influences, and peer influences subscales of the Psychosocial Constructs for Adolescent Physical Activity and Sedentary Behaviors | 5 months
  Social motivation will be assessed using the decisional balance, family influences, and peer influences subscales
Participants' self-efficacy for diet will be assessed using the Psychosocial Constructs for Adolescent Fruit and Vegetables and Dietary Fat Intake | 5 months
  Self-efficacy beliefs related to diet
Participants' self-efficacy for physical activity will be assessed using the Psychosocial Constructs for Adolescent Physical Activity and Sedentary Behaviors | 5 months
  Self efficacy beliefs related to behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Sasha A Fleary, PhD, Principal Investigator — City University of New York
Locations (1):
- Neighborhood House Charter School, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fleary SA. A Web-Based Intervention to Improve Health Literacy and Obesogenic Behaviors Among Adolescents: Protocol of a Randomized Pilot Feasibility Study for a Parallel Randomized Controlled Trial. JMIR Res Protoc. 2022 Aug 16;11(8):e40191. doi: 10.2196/40191. PMID 35972787